CLINICAL TRIAL: NCT00803244
Title: A Randomised, Double-blind, Placebo-controlled, Multi National, Phase III Study of the Efficacy and Safety of 300 IR Sublingual Immunotherapy (SLIT) Tablet, Starting 2 Months Before the Grass Pollen Season Once Daily to Patients Suffering From Grass Pollen Rhinoconjunctivitis
Brief Title: Safety and Efficacy on Phase III Study on 300 IR SLIT to Patients Suffering From Grass Pollen Rhinoconjunctivitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Stallergenes Greer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VO60.08
Record Dates: First submitted 2008-11-27; First posted 2008-12-05 (Estimated); Results first posted 2016-05-25 (Estimated); Last update posted 2016-05-25 (Estimated); Status verified 2016-04

CONDITIONS: Primary Disease
Keywords: allergic rhinoconjunctivitis
MeSH Terms: interventions — Sublingual Immunotherapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 300 IR (Experimental): 300 IR grass pollen allergen extract tablet
  Interventions: Drug: 300 IR
- Placebo (Placebo Comparator): Placebo tablet
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: 300 IR — 300 IR grass pollen allergen extract tablet starting 2 months before the grass pollen season and during the grass pollen season
  Other Names: Sublingual immunotherapy tablet
  Arms: 300 IR
Drug: Placebo — Placebo sublingual tablet starting 2 months before the grass pollen season and during the grass pollen season
  Other Names: Sublingual placebo tablet
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of sublingual tablets of grass pollen allergen extract when initiated 2 months before the grass pollen season compared with placebo for reduction of rhinoconjunctivitis symptoms and rescue medication usage.

DETAILED DESCRIPTION:
To assess the efficacy of sublingual tablets of grass pollen allergen extract when initiated 2 months before the grass pollen season on:

- The Average Adjusted Symptom Score (AASS).

To document the safety of the treatment.

ELIGIBILITY:
Inclusion criteria:

1. Male or female outpatients aged 12 to 65 years (inclusive).
2. Patients with grass pollen-related allergic rhinoconjunctivitis for at least the last two grass pollen seasons.
3. Positive SPT
4. RRTSS during the previous pollen season of greater than or equal to 12 out of a possible 18.

Exclusion Criteria:

1. Positive SPT to any other seasonal allergens present during the grass pollen season
2. Patients with clinically significant confounding symptoms of allergy to other allergens
3. Significant symptomatic perennial allergy due to an allergen to which the patient is regularly exposed.
4. Patients with moderate or severe persistent asthma (Global Initiative for Asthma [GINA] 3 or 4).

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 381 (Actual)
Dates: Start 2009-01; Primary Completion 2009-08 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: DE BLAY Frédéric, MD, Principal Investigator — NHC, Hôpitaux Universitaires de Strasbourg
Locations (6):
- France (3):
  - Stallergenes Sa, Antony
  - Hop Montauban, Montauban
  - Cab medical, Orange
- Azienda Ospedaliera, Parma, Italy
- Spain (2):
  - Complejo Hospitalario de Caceres, Cáceres
  - HGU La Paz, Madrid

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First Patient First Visit 28 JAN 2009, Last Patient Last Visit 31 AUG 2009
Period: Overall Study
Arm/Group | 300 IR | Placebo
Started | 188 | 193
Completed | 181 | 178
Not Completed | 7 | 15
Not completed — Adverse Event | 1 | 2
Not completed — Withdrawal by Subject | 2 | 3
Not completed — Any other reason not above-mentioned | 4 | 10

BASELINE CHARACTERISTICS:
Population: Safety Set: The Safety Set included all patients who received at least one dose of the investigational product.
  The Full Analysis Set included all patients who received at least one dose of the investigational product and had at least one Adjusted Symptom Score during the pollen period while on treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | 300 IR | Placebo | Total
Number analyzed (Participants) | 178 | 185 | 363
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.5 (10.53) | 29.6 (9.87) | 30.0 (10.20)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 77 | 79 | 156
  Male | 101 | 106 | 207

OUTCOME MEASURES:

1. Primary Outcome: Average Adjusted Symptom Score (AAdSS)
Description: The Adjusted Symptom Score (AdSS) is a subject-specific symptom score which is adjusted for rescue medication use.
  Participants assessed daily, during the pollen period while on treatment, 6 rhinoconjunctivitis symptoms (sneezing, rhinorrhea, nasal pruritus, nasal congestion, ocular pruritus and watery eyes) each symptom is scored as follows: 0: no symptoms, 1: mild symptoms, 2: moderate symptoms, 3: severe symptoms. The sum of the 6 symptoms is the Rhinoconjunctivitis Total Symptom Score (RTSS) (range 0-18). If the subject took rescue medication on a given day, the AdSS equals the RTSS of that day or the AdSS of the day before, whichever is higher. This adjustment applies to the day of rescue medication use and the following day. Like the RTSS, the AdSS ranges from 0 to 18. The lower the score, the better the outcome.
Time Frame: Pollen period (average of 32.1 days)
Population: The Full Analysis Set included all patients who received at least one dose of the investigational product and had at least one Adjusted Symptom Score during the pollen period while on treatment.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale (range: 0 to 18)
Arm/Group | 300 IR | Placebo
Number analyzed (Participants) | 178 | 184
Units on a scale (range: 0 to 18) | 5.58 (0.330) | 6.07 (0.335)
Statistical Analysis 1: Comparison: 300 IR vs Placebo; Test type: Superiority or Other; p = 0.2344, ANCOVA; Difference in LS Means = -0.49, 95% CI [-1.30 to 0.32]

2. Post Hoc Outcome: Combined Score (CS)
Description: The daily Combined Score (CS) is a patient specific score taking into account the patient's daily Rhinoconjunctivis Total Symptom Score (RTSS) and daily Rescue Medication Score (RMS), assuming equivalent importance of symptoms and rescue medication scores.
  The RMS (range 0-3) is derived as follows: 0, no rescue medication; 1, use of antihistamine; 2, use of nasal corticosteroid; 3, use of oral corticosteroid. The RTSS (range 0-18) is the sum of the 6 individual rhinoconjunctivitis symptom score (each symptom is scored as follows: 0: no symptoms, 1: mild symptoms, 2: moderate symptoms and 3: severe symptoms).
  The CS (range 0-3) = (RTSS/6 + RMS)/2. The lower the score, the better the outcome.
Time Frame: Pollen period (average of 32.1 days)
Population: The Full Analysis Set included all patients who received at least one dose of the investigational product and had at least one Combined Score during the pollen period while on treatment.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale (range: 0 to 3)
Arm/Group | 300 IR | Placebo
Number analyzed (Participants) | 178 | 182
Units on a scale (range: 0 to 3) | 0.38 (0.038) | 0.48 (0.038)
Statistical Analysis 1: Comparison: 300 IR vs Placebo; Test type: Superiority or Other; p = 0.0401, ANCOVA; LS Mean difference vs. Placebo = -0.09, 95% CI 2-sided [-0.18 to 0.00] — Relative LS Means difference (%) = -19.7

ADVERSE EVENTS:
Time Frame: 2 months before the pollen period until the end of the pollen period.
Description: A treatment-emergent adverse event (TEAE) is defined as any AE that started on or after the first dose of the investigational product was administered and is ongoing, or ended on or after the first dose of the investigational product.
Arm/Group | 300 IR | Placebo
Serious Adverse Events (participants affected / at risk) | 1/188 | 1/193
Other Adverse Events (participants affected / at risk) | 110/188 | 63/193
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 300 IR (N=188) | Placebo (N=193)
JOINT DISLOCATION (Injury, poisoning and procedural complications) | 0 | 1
TIBIA FRACTURE (Injury, poisoning and procedural complications) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 300 IR (N=188) | Placebo (N=193)
ORAL PRURITUS (Gastrointestinal disorders) | 60 | 5
OEDEMA MOUTH (Gastrointestinal disorders) | 13 | 0
THROAT IRRITATION (Respiratory, thoracic and mediastinal disorders) | 31 | 9
COUGH (Respiratory, thoracic and mediastinal disorders) | 9 | 11
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 8 | 12
HEADACHE (Nervous system disorders) | 32 | 32
NASOPHARYNGITIS (Infections and infestations) | 11 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No